CLINICAL TRIAL: NCT04267302
Title: Baby Item Learning and Development Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20190970
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Infant Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baby Bouncer Group (Other): Participants in the group will be receiving a baby bouncer for use from infant's birth up to 8 months after birth.
  Interventions: Other: Baby Bouncer
- Baby Bouncer Group with Infant T-Shirt with LENA (Other): A subsample of the participants in the baby bouncer group will also receive infant t-shirts with wearable audio recorders.
  Interventions: Other: Baby Bouncer; Other: Infant t-shirts with Language Environment Analysis (LENA) audio recorders
- Baby Carrier Group (Other): Participants in the group will be receiving a baby carrier for use from infant's birth up to 8 months after birth.
  Interventions: Other: Baby Carrier
- Baby Carrier Group with Infant T-Shirt with LENA (Other): A subsample of the participants in the baby carrier group will also receive infant t-shirts with wearable audio recorders.
  Interventions: Other: Infant t-shirts with Language Environment Analysis (LENA) audio recorders; Other: Baby Carrier

INTERVENTIONS:
Other: Baby Bouncer — Fischer Price baby bouncer.
  Arms: Baby Bouncer Group; Baby Bouncer Group with Infant T-Shirt with LENA
Other: Infant t-shirts with Language Environment Analysis (LENA) audio recorders — Infant t-shirts with wearable LENA audio recorders for 2-8 hours of recordings of vocal interaction, crying and turn-taking.
  Arms: Baby Bouncer Group with Infant T-Shirt with LENA; Baby Carrier Group with Infant T-Shirt with LENA
Other: Baby Carrier — Ergobaby Baby carrier.
  Arms: Baby Carrier Group; Baby Carrier Group with Infant T-Shirt with LENA

SUMMARY:
The goal of this study is to experimentally test whether baby items can promote healthy infant development.

ELIGIBILITY:
Inclusion Criteria:

* Mothers and their infants must be healthy with no known birth complications
* Infants must be born full term (at least 37 weeks gestation)
* Mother must speak English
* Mothers must be at least 28 weeks along in their pregnancy. Mothers with newborns who are less than 2 weeks will be included.

Exclusion Criteria:

* Participants who does not meet all the inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive skill as assessed via eye tracking | 8 months
  Cognitive skill is reported as the percentage of accuracy of eye gaze as evaluated via the eye tracking procedure.
Parental Engagement | 8 months
  Mother and infant will engage in a 15-minute unstructured free playtime. This engagement will be videotaped and assessed by the Investigator. Parental engagement is reported as the percentage of parental sensitivity and synchrony scored on a 0-100% scale with the higher score indicating increased sensitivity and synchrony.
Infant Reactivity (Crying) assessed by the Face to Face/Still Face Procedure | 8 months
  Infant emotions and social engagement is reported as the time noted when the infant was crying during the 6 minute Face to Face/Still Face Procedure.
Infant Reactivity (Smiling) assessed by the Face to Face/Still Face Procedure | 8 months
  Infant emotions and social engagement is reported as the time noted when the infant was smiling during the 6 minute Face to Face/Still Face Procedure.
Oxytocin levels | 8 months
  Mother and infant oxytocin levels will be measured via saliva sample.
Percentage of infant and adult vocalizations time | Up to 8 hours
  Assessed via 2-8 hours audio recordings on LENA.
Percentage of infant and adult turn taking | Up to 8 hours
  Assessed via 2-8 hours audio recordings on LENA. Turn taking is defined as the verbal exchange by adult and infant.
Percentage of Infant crying time | Up to 8 hours
  Percentage of infant crying time will be assessed via 2-8 hours audio recordings on LENA.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Simpson, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No